CLINICAL TRIAL: NCT03166904
Title: AZD2014 in RICTOR Amplified Solid Cancer
Brief Title: Phase II Trial of AZD2014 in RICTOR Amplified Solid Cancer Patients Refractory to Standard Chemotherapy
Acronym: RICTOR_SC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-05-097
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — vistusertib

STUDY DESIGN:
Intervention Model Description: Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD2014 (Experimental): Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle
  Interventions: Drug: Vistusertib(AZD2014)

INTERVENTIONS:
Drug: Vistusertib(AZD2014) — Vistusertib(AZD2014) is a selective dual mTOR kinase inhibitor targeting both mTORC1 (rapamycin sensitive) and mTORC2 (rapamycin insensitive) complexes of mammalian Target Of Rapamycin (mTOR).
  Other Names: azd2014

SUMMARY:
Patients with RICTOR amplified refractory solid cancer will receive vistusertib(AZD2014). Study-arm is composed of 27 patients.

Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date of first dose, up to week 40, then every 16 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

DETAILED DESCRIPTION:
Patients with RICTOR amplified refractory solid cancer will receive vistusertib(AZD2014). Study-arm is composed of 27 patients.

Vistusertib(AZD2014) 50mg BD continuous schedule of a 28 day cycle Tumour evaluation using RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date of first dose, up to week 40, then every 16 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

Study treatment will be continued until objective disease progression (unless other criteria for treatment discontinuation are met). Patients may continue vistusertib(AZD2014) beyond progression (according to RECIST 1.1), at the discretion of the investigator if they are clinically benefiting from the treatment and they do not meet any other discontinuation criteria.

If a patient discontinues study treatment prior to disease progression, they should continue to be assessed using RECIST 1.1 until disease progression and then followed up for survival.

Assessments for survival should be made every 8 weeks following objective disease progression. The details of first and subsequent therapies for cancer, after discontinuation of treatment, will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid cancers (including histologically or cytologically documented gastric cancer, colorectal cancer, hepatoma, biliary tract cancers, pancreatic cancer and rare cancers.) that has progressed after standard chemotherapy.

   - Rare cancers are defined as sarcoma, neuroendocrine carcinoma
2. Provision of tumor sample tumor sample tumor sample tumor sampletumor sample (from either a resection or biopsy)
3. Patients with RICTOR amplification through NGS.
4. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. Patients not having received recommended treatment-lines and chemotherapy regimen for the treatment of each tumor type in the advanced setting.
2. Any previous treatment with PIK3CA, AKT or mTOR inhibitor or agents with mixed PI3K / mTOR activity.
3. HER2 positive AGC patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Objective reponse rate (ORR) by RECIST 1.1 | 12months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea